CLINICAL TRIAL: NCT06076447
Title: Cross-Cultural Adaptation and Validation of the Urdu Version of the Minnesota Living With Heart Failure Questionnaire (MLHFQ) Among Individuals With Heart Failure
Brief Title: Urdu Translation and Validation of MLHFQ
Status: Recruiting | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/PhD/01199 Iqbal Project B
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* To translate the Minnesota Living with Heart Failure Questionnaire (MLHFQ) questionnaire into Urdu language of Pakistan.
* To determine the validity and reliability of cross cultural adapted and Urdu translated MLHFQ questionnaire version among HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure who sought treatment at the outpatient cardiology clinic.
* Who could read and write in Urdu and English language and are willing to participate in the study.

Exclusion Criteria:

* Decline consent
* Communication barriers or cognitive disorder as well as those with exacerbated condition and those who were not available for re-test were excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Heart Failure individuals
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-11-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life (Minnesota Living with Heart Failure Questionnaire) | 6 months
  Quality of life will be measured through Minnesota Living with Heart Failure Questionnaire (MLHFQ). It is one of the most widely used health-related quality of life questionnaires for individuals with HF. It provides scores for two dimensions, physical and emotional, and a total score. The MLHFQ is a self-administered, 21-item disease-specific instrument for individuals with HF. Each item is scored in a 6-point Likert Scale (0 to 5), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life. The MLHFQ has two domains; physical domain (eight items, score range from 0 to 40) and emotional domain (five items, score range from 0 to 25).

SECONDARY OUTCOMES:
Reliability of translated versions of Minnesota Living with Heart Failure Questionnaire | 6 months
  To determine reliability of MLHFQ in (URDU) language. Reliability refers to ability of a measure to produce same results administered at two or more intervals. Thus this will be test through test retest reliability
Validity of translated versions of Minnesota Living with Heart Failure Questionnaire | 6 months
  To determine the validity of translation of MLHFQ. in (URDU) language. Validity is defined as how accurate the results are. Thus this will be measured through various parameters

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University; Arshad Nawaz Malik, PhD, Study Chair — Riphah International University; Shane Patman, PhD, Study Chair — University of Notre Dame Australia
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No